CLINICAL TRIAL: NCT01195025
Title: Volume Kinetics for Starch Solution and Acetated Ringers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Joachim Zdolsek, MD, PhD, University Hospital, Linkoeping
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VkVR
Record Dates: First submitted 2010-08-31; First posted 2010-09-03 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Blood Volume; Blood Coagulation
Keywords: Blood volume; blood coagulation; volume kinetics
MeSH Terms: conditions — Thrombosis | interventions — Colloids; HES 130-0.4

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- A.acetatedRingers, B.colloid & C.colloid+acetatedRingers (Other): First intervention: A. acetated Ringers 20 ml/kg bodyweight during 30 minutes followed by 150 minutes of equilibration, when blood samples were collected.
  Washout >7 days
  Second intervention: B. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed by 390 minutes of equilibration and blood samples.
  Washout > 7 Days
  Third intervention: C. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed 90 minutes later by acetated Ringers 20 ml/kg bodyweight during 30 minutes. thereafter the subjects stayed for Another 285 minutes of equilibration and blood samples.
  Interventions: Drug: acetated Ringers; Drug: colloid; Drug: colloid+acetated Ringer; Device: Non-invasive hemoglobin with pulse-oximeter (SpHb)
- A.colloid, B.colloid+acetatedRinger & C.acetatedRingers (Other): First intervention: A. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed by 390 minutes of equilibration and blood samples.
  Washout >7 days
  Second intervention: B. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed 90 minutes later by acetated Ringers 20 ml/kg bodyweight during 30 minutes. thereafter the subjects stayed for Another 285 minutes of equilibration and blood samples.
  Washout > 7 Days
  Third intervention: C. acetated Ringers 20 ml/kg bodyweight during 30 minutes followed by150 minutes of equilibration, when blood samples were collected.
  Interventions: Drug: acetated Ringers; Drug: colloid; Drug: colloid+acetated Ringer; Device: Non-invasive hemoglobin with pulse-oximeter (SpHb)
- A.acetatedRingers, B.acetatedRingers+colloid & C.colloid (Other): First intervention: A. acetated Ringers 20 ml/kg bodyweight during 30 minutes followed by150 minutes of equilibration, when blood samples were collected.
  Washout >7 days
  Second intervention: B.Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed 90 minutes later by acetated Ringers 20 ml/kg bodyweight during 30 minutes. thereafter the subjects stayed for Another 285 minutes of equilibration and blood samples.
  Washout > 7 Days
  Third intervention: C. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed by 390 minutes of equilibration and blood samples.
  Interventions: Drug: acetated Ringers; Drug: colloid; Drug: colloid+acetated Ringer; Device: Non-invasive hemoglobin with pulse-oximeter (SpHb)
- A.colloid, B.acetatedRingers & C.colloid+acetatedRingers (Other): First intervention: A. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed by 390 minutes of equilibration and blood samples.acetated Ringers 20 ml/kg bodyweight during 30 minutes followed by150 minutes of equilibration, when blood samples were collected.
  Washout >7 days
  Second intervention: B. acetated Ringers 20 ml/kg bodyweight during 30 minutes followed by150 minutes of equilibration, when blood samples were collected.
  Washout > 7 Days
  Third intervention: C. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed 90 minutes later by acetated Ringers 20 ml/kg bodyweight during 30 minutes. thereafter the subjects stayed for Another 285 minutes of equilibration and blood samples.
  Interventions: Drug: acetated Ringers; Drug: colloid; Drug: colloid+acetated Ringer; Device: Non-invasive hemoglobin with pulse-oximeter (SpHb)
- A.colloid+acetatedRingers, B.colloid & C.acetated Ringers (Other): First intervention: A. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed 90 minutes later by acetated Ringers 20 ml/kg bodyweight during 30 minutes. thereafter the subjects stayed for Another 285 minutes of equilibration and blood samples.
  Washout >7 days
  Second intervention: B. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed by 390 minutes of equilibration and blood samples.
  Washout > 7 Days
  Third intervention: C. acetated Ringers 20 ml/kg bodyweight during 30 minutes followed by150 minutes of equilibration, when blood samples were collected.
  Interventions: Drug: acetated Ringers; Drug: colloid; Drug: colloid+acetated Ringer; Device: Non-invasive hemoglobin with pulse-oximeter (SpHb)

INTERVENTIONS:
Drug: acetated Ringers — Infusion of Ringer acetate 20 ml/kg over 30 min
Drug: colloid — Infusion of starch 10 ml/kg over 30 min
  Other Names: Voluven
Drug: colloid+acetated Ringer — Infusion of combined colloid+acetated Ringer; 10 ml/kg of starch was infused between 0 and 30 min, followed by 20 ml/kg of Ringers acetate between 105 and 135 min.
  Other Names: Voluven; acetated Ringers
Device: Non-invasive hemoglobin with pulse-oximeter (SpHb) — Non-invasive hemoglobin with pulse-oximeter (SpHb) was measured in all subjects, during all infusions.
  Other Names: Radical 7, Masimo

SUMMARY:
Volume kinetics is a method mostly used, so far, to study the distribution and elimination of crystalloid solutions. Voluven (in Sweden the most commonly used colloid for replacement of bleeding during surgery) is poorly studied, though. Also, a recent study showed unexpected volume kinetics for a crystalloid solution when it was given after a colloid solution. The investigators aim to study the volume kinetics of crystalloids and colloids and also the combination of the two in more detail. The investigators will also compare the invasive hemoglobin measurements with measurements from a new non-invasive tool (Radical 7, from Masimo Inc.) which could help to make volume kinetics more practical for everyday use. Finally the investigators will also study the concentrations of a few coagulation factors to see if they can explain the variations in coagulability that has been described in earlier studies of infusion solutions.

DETAILED DESCRIPTION:
We will study ten volunteers, each one on three occasions. Each volunteer will receive only crystalloid one time, only colloid another time, and on the third occasion first a colloid and then a crystalloid one hour later. The different protocols will be in random order in the different volunteers. During all these tests we will sample the hemoglobin (both invasive and non-invasive) every fifth minute in the beginning (every tenth minute later) after the infusion. On six to nine occasions during each test we will analyse Albumin, Cystatin-C, Ig-G, Ig-M as markers of hemodilution and D-Dimer, Fibrinogen, Factor VII, PK-INR (prothrombin complex international normalized ratio), and aPTT (activated partial thromboplastin time) as markers of coagulation. The volunteers are also monitored regarding non-invasive blood pressure and pulse rate.

ELIGIBILITY:
Inclusion Criteria: healthy males between 20 and 50 years were advertised for. Males due to simplified urine collection during supine position.

Exclusion Criteria:

under age < 18 years

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Zdolsek, MD, PhD, Principal Investigator — University Hospital, Linköping, Sweden
Locations (1):
- University Hospital, Intensive care unit, Linköping, Linköping, Sweden

REFERENCES:
- [Derived] Hahn RG, Wuethrich PY, Zdolsek JH. Can perioperative hemodilution be monitored with non-invasive measurement of blood hemoglobin? BMC Anesthesiol. 2021 May 6;21(1):138. doi: 10.1186/s12871-021-01351-4. PMID 33957864
- [Derived] Hahn RG, Bergek C, Geback T, Zdolsek J. Interactions between the volume effects of hydroxyethyl starch 130/0.4 and Ringer s acetate. Crit Care. 2013 May 29;17(3):R104. doi: 10.1186/cc12749. PMID 23718743
- [Derived] Bergek C, Zdolsek JH, Hahn RG. Accuracy of noninvasive haemoglobin measurement by pulse oximetry depends on the type of infusion fluid. Eur J Anaesthesiol. 2013 Feb;30(2):73-9. doi: 10.1097/EJA.0b013e3283592733. PMID 23303244 (Retraction: PMID 24887135 Eur J Anaesthesiol. 2014 Jul;31(7):396)
- [Derived] Bergek C, Zdolsek JH, Hahn RG. Accuracy of noninvasive haemoglobin measurement by pulse oximetry depends on the type of infusion fluid. Eur J Anaesthesiol. 2012 Dec;29(12):586-92. doi: 10.1097/EJA.0b013e3283592733. PMID 23047301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 Healthy male volunteers 18 to 50 years old
Pre-assignment Details: Random crossover study, with at least one week between every study occasion.
Groups:
- A. Acetated Ringers, B.Colloid and C. Colloid+Acetated Ringers: First intervention: A. acetated Ringers 20 ml/kg bodyweight during 30 minutes followed by150 minutes of equilibration, when blood samples were collected.
  Washout >7 days
  Second intervention: B. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed by 390 minutes of equilibration and blood samples.
  Washout > 7 Days
  Third intervention: C. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed 90 minutes later by acetated Ringers 20 ml/kg bodyweight during 30 minutes. thereafter the subjects stayed for Another 285 minutes of equilibration and blood samples.
- A. Colloid, B. Colloid+Acetated Ringers and C.Acetated Ringers: First intervention: A. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed by 390 minutes of equilibration and blood samples.
  Washout >7 days
  Second intervention: B. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed 90 minutes later by acetated Ringers 20 ml/kg bodyweight during 30 minutes. thereafter the subjects stayed for Another 285 minutes of equilibration and blood samples.
  Washout > 7 Days
  Third intervention: C. acetated Ringers 20 ml/kg bodyweight during 30 minutes followed by150 minutes of equilibration, when blood samples were collected
- A. Acetated Ringers, B. Colloid+Acetated Ringers and C.Colloid: First intervention: A. acetated Ringers 20 ml/kg bodyweight during 30 minutes followed by 150 minutes of equilibration, when blood samples were collected
  Washout >7 days
  Second intervention: B. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed 90 minutes later by acetated Ringers 20 ml/kg bodyweight during 30 minutes. thereafter the subjects stayed for Another 285 minutes of equilibration and blood samples.
  Washout > 7 Days
  Third intervention: C. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed by 390 minutes of equilibration and blood samples.
- A.Colloid, B. Acetated Ringers and C. Colloid+Acetated Ringers: First intervention: A. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed by 390 minutes of equilibration and blood samples.
  Washout >7 days
  Second intervention: B. acetated Ringers 20 ml/kg bodyweight during 30 minutes followed by150 minutes of equilibration, when blood samples were collected.
  Washout > 7 Days
  Third intervention: C. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed 90 minutes later by acetated Ringers 20 ml/kg bodyweight during 30 minutes. thereafter the subjects stayed for Another 285 minutes of equilibration and blood samples.
- A. Colloid+Acetated Ringers, B.Colloid and C. Acetated Ringers: First intervention: A. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed 90 minutes later by acetated Ringers 20 ml/kg bodyweight during 30 minutes. thereafter the subjects stayed for Another 285 minutes of equilibration and blood samples.
  Washout >7 days
  Second intervention: B. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed by 390 minutes of equilibration and blood samples.
  Washout > 7 Days
  Third intervention: C. acetated Ringers 20 ml/kg bodyweight during 30 minutes followed by150 minutes of equilibration, when blood samples were collected.
Period: First Intervention A
Arm/Group | A. Acetated Ringers, B.Colloid and C. Colloid+Acetated Ringers | A. Colloid, B. Colloid+Acetated Ringers and C.Acetated Ringers | A. Acetated Ringers, B. Colloid+Acetated Ringers and C.Colloid | A.Colloid, B. Acetated Ringers and C. Colloid+Acetated Ringers | A. Colloid+Acetated Ringers, B.Colloid and C. Acetated Ringers
Started | 2 | 3 | 2 | 2 | 1
Completed | 2 | 3 | 2 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Second Intervention B
Arm/Group | A. Acetated Ringers, B.Colloid and C. Colloid+Acetated Ringers | A. Colloid, B. Colloid+Acetated Ringers and C.Acetated Ringers | A. Acetated Ringers, B. Colloid+Acetated Ringers and C.Colloid | A.Colloid, B. Acetated Ringers and C. Colloid+Acetated Ringers | A. Colloid+Acetated Ringers, B.Colloid and C. Acetated Ringers
Started | 2 | 3 | 2 | 2 | 1
Completed | 2 | 3 | 2 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Third Intervention C
Arm/Group | A. Acetated Ringers, B.Colloid and C. Colloid+Acetated Ringers | A. Colloid, B. Colloid+Acetated Ringers and C.Acetated Ringers | A. Acetated Ringers, B. Colloid+Acetated Ringers and C.Colloid | A.Colloid, B. Acetated Ringers and C. Colloid+Acetated Ringers | A. Colloid+Acetated Ringers, B.Colloid and C. Acetated Ringers
Started | 2 | 3 | 2 | 2 | 1
Completed | 2 | 3 | 2 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dilution Effects of iv Fluids: Three experiments:
  A. acetated Ringers 20 ml/kg bodyweight during 30 minutes B. Hydroxy ethyl starch (HES) 6% 10 mL/kg bodyweight during 30 min C. A combination of A and B. HES during 0-30 min and Ringer's during 105-135 minutes.
Arm/Group | Dilution Effects of iv Fluids
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  Sweden | 10

OUTCOME MEASURES:

1. Primary Outcome: Volume Effects for Hydroxyethyl Starch, Ringer's Solution or a Combination of Both.
Description: volume kinetics: mathematical calculation from hemoglobin variations during and after an infusion.
  Degree of plasma dilution depending on which solution(s) and how much solution is/are given.
Time Frame: 420 minutes
Population: All the 10 participating subjects. Analysis studying the summary of each of the included infusion occasions. Only acetated Ringers, only colloid and finally a combination of colloid and acetated Ringers.
  Each experiment generated one distribution volume. (In experiment C one for acetated Ringer's and one for Starch (HES 6%)).
Measure: Median (Inter-Quartile Range); unit: Litre
Groups:
- Hydroxyethyl Starch, Ringers and a Combination of Both.: A. acetated Ringers 20 ml/kg bodyweight during 30 minutes B. Hydroxyethyl starch (HES 6 %, 10 ml/kg bodyweight during 30 minutes. C. Hydroxyethyl starch (HES 6 %, 10 ml/kg bodyweight during 30 minutes followed 90 minutes later by acetated Ringers 20 ml/kg bodyweight during 30 minutes.
Arm/Group | Hydroxyethyl Starch, Ringers and a Combination of Both.
Number analyzed (Participants) | 10
Litre
  Distribution volume of Acetated Ringers | 5.53 [4.25 to 7.31]
  Distribution volume for HES 6% | 2.94 [2.65 to 3.31]
  Distribution vol for HES combined with Ringer's | 3.12 [3.01 to 3.45]
  Distribution vol for Ringers combined with HES | 4 [3.05 to 4.82]

2. Secondary Outcome: Accuracy of Non-invasive Hemoglobin Monitoring for Different Fluids
Description: Pulse-oximeter based measurements compared with invasive hemoglobin measurements. All paired in the study.
  Accuracy depending on which infusion is selected (Ringer's, Hydroxyethyl starch or a combination of both).
Time Frame: 420 min
Population: The study was analysed per protocol and missing values were not replaced. All pairs of all collected data in one series of experiments. The number of analysed data points for each subject was in experiment A: 26, in experiment B: 32 and in experiment C: 42.
Measure: Median (Inter-Quartile Range); unit: percentage of relative difference
Units Other Than Participants: Hemoglobin measurements (pairs)
Groups:
- Venous Hemoglobin and Non-invasive Hemoglobin (SpHb): A comparison of all paired hemoglobin measurements (B-Hb and SpHb) during the experiments for all the 10 volunteers.
  Relative difference(%) = (SpHb - Hb)/((Hb+SpHb)/2) x 100
Arm/Group | Venous Hemoglobin and Non-invasive Hemoglobin (SpHb)
Number analyzed (Participants) | 10
Number analyzed (Hemoglobin measurements (pairs)) | 956
percentage of relative difference
  Ringers acetate | -5.3 [-10.4 to 1.5]
  HES 6% | 0.0 [-6.8 to 4.6]
  HES 6% + Ringers acetate | 1.5 [-4.9 to 10.9]

3. Secondary Outcome: Accuracy of Noninvasive Haemoglobin Measurement by Pulse Oximetry, for Different Fluids (Start to End of Infusion)
Description: Difference between true hemoglobin B-Hb and measured hemoglobin with pulseoximeter (SpHb)at the end of an infusion in relation to the initial measured values SpHb and B-Hb at the start of the infusion.
  Relative difference (%) = (SpHb - Hb)/((Hb+SpHb)/2) x 100
Time Frame: 30 min
Population: Only the pure experiments were included in this analysis. The combined experiment is not included since infusions were performed in sequence, which made the comparison of the bias for the two different fluids irrelevant.
Measure: Median (Inter-Quartile Range); unit: percentage of relative difference
Units Other Than Participants: SpHb - B-Hgb
Groups:
- Colloid (Voluven), Acetated Ringers and a Combination of Both.: A. acetated Ringers 20 ml/kg bodyweight during 30 minutes B. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes
  The combined experiment is not included since infusions were performed in sequence, which made the comparison of the bias for the two different fluids irrelevant.
Arm/Group | Colloid (Voluven), Acetated Ringers and a Combination of Both.
Number analyzed (Participants) | 10
Number analyzed (SpHb - B-Hgb) | 20
percentage of relative difference
  Ringer's acetate | 7 [2.5 to 11.1]
  Hydroxy ethyl starch 6% | -4.3 [-7.2 to -0.9]

4. Secondary Outcome: Variation of Coagulation Factors and Plasma Proteins During and After Infusion of Crystalloid and Colloid Solutions.
Description: The investigators will measure a few markers of coagulation (fibrinogen, thrombocytes, D-Dimer, PK-INR, aPTT, and coagulation factor VII) as well as Cystatin C, serum albumine and hemoglobin and how the concentration of these vary with the different dilutions of blood during and after infusion of a colloid and/or a crystalloid solution.
Time Frame: 420 minutes
Reporting Status: Not Posted, anticipated posting 2015-05

5. Primary Outcome: Elimination Half Life for Different Fluids Alone or When Combined
Description: Volume kinetic analyses of the dilution of hemoglobin for different infusion fluids alone or in combination.
Time Frame: 420 minutes
Population: All the 10 participating subjects. Analysis studying the summary of each of the included infusion occasions. Only acetated Ringers, only colloid and finally a combination of colloid and acetated Ringers. Each experiment generated one elimination half-life (In experiment C one for acetated Ringer's and one for starch (HES 6%)).
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Infusion protocols
Arm/Group | Hydroxyethyl Starch, Ringers and a Combination of Both.
Number analyzed (Participants) | 10
Number analyzed (Infusion protocols) | 30
Minutes
  Elimination half life for Ringer's | 88 [54 to 150]
  Elimination half life for HES | 116 [87 to 152]
  Elimination half life for HES (+ Ringer's) | 126 [75 to 150]
  Elimination half life for Ringer's (+ HES) | 497 [146 to 805]

ADVERSE EVENTS:
Groups:
- Colloid-, Acetated Ringers and Combined: Voluven, acetated Ringers: Infusions at three different occasions separated by at least one week.
  A. acetated Ringers 25 ml/kg bodyweight during 30 minutes B. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes. C. Voluven 6 % (starch solution) 10 ml/kg bodyweight during 30 minutes followed 90 minutes later by acetated Ringers 15 ml/kg bodyweight during 30 minutes.
Arm/Group | Colloid-, Acetated Ringers and Combined
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes